CLINICAL TRIAL: NCT06354010
Title: Cross-sectional and Prospective Study to Characterize Early-onset Presbycusis
Acronym: SONG
Status: Recruiting | Type: Observational
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Other Study IDs: SENS-NH02
Record Dates: First submitted 2024-02-20; First posted 2024-04-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: Adulthood-onset bilateral sensorineural hearing loss; GJB2; Presbycusis; hearing impairement; Deafness; Connexin 26; SONG; Genetic deafness; Adult deafness
MeSH Terms: conditions — Hearing Loss, Sensorineural; Presbycusis; Deafness | interventions — Genotype

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with adulthood-onset bilateral sensorineural hearing loss (SNHL)
  Interventions: Genetic: Genotyping
- Patients that carry mutations in the gene GJB2 from patients with adulthood-onset bilateral SNHL
  Interventions: Other: Audiological assessments

INTERVENTIONS:
Genetic: Genotyping — Genotyping to determine if patients present mutations to the gene GJB2.
  Groups: Patients with adulthood-onset bilateral sensorineural hearing loss (SNHL)
Other: Audiological assessments — Audiological assessments
  Groups: Patients that carry mutations in the gene GJB2 from patients with adulthood-onset bilateral SNHL

SUMMARY:
The purpose of this study is to characterize and assess the evolution of hearing impairment of patients with adulthood-onset bilateral sensorineural hearing loss carrying mutations on GJB2 gene.

DETAILED DESCRIPTION:
This study aims to characterize patients with adulthood-onset bilateral sensorineural hearing loss not due to any underlying medical condition (likely due to a genetic cause) and to assess the evolution of hearing impairment of those carrying mutations in GJB2 gene.

Patients who present with adulthood-onset bilateral sensorineural hearing loss will be screened for the presence of mutation involved in hearing impairment. Patients with GJB2 mutations will be proposed to continue in a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients ≥30 and ≤55 years old
2. Bilateral hearing loss first noticed after the age of 16 years old
3. Documented genotyping results showing mutations in GJB2 gene.

Exclusion Criteria:

1. Deafness with a known, non-genetic cause
2. To the opinion of the investigator, unable and/or unwilling to comply with all the protocol requirements and/or study procedures

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female participants aged ≥30 and ≤55 years old with bilateral hearing loss first noticed after the age of 16 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of hearing impairment of adult patients with early-onset presbycusis carrying mutations in GJB2 gene. | 2 years
  Evolution of hearing impairment assessed by Pure Tone Audiometry
Evolution of hearing impairment of adult patients with early-onset presbycusis carrying mutations in GJB2 gene | 2 years
  Evolution of hearing impairment assessed by Speech in noise

SECONDARY OUTCOMES:
Genetic characteristics of adult patients with early-onset presbycusis | Unique visit
  Genotyping
Audiological characteristics of adult patients with early-onset presbycusis | Unique visit
  Pure Tone Audiometry
Mood evaluation in adult patients with early-onset presbycusis carrying mutations in GJB2 gene | 2 years
  Mood evaluation assessed with Patient Health Questionnaire for depression (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Venail, Pr, Principal Investigator — CHU Montpellier - Hôpital Gui de Chauliac
Locations (2):
- The University of South Florida Board of Trustees, Tampa, Florida, United States
- CHU Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No